CLINICAL TRIAL: NCT06796556
Title: Evaluation of an Algorithm for the Identification of Post-traumatic Stress Disorder
Acronym: Dstress
Status: Completed | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A02717-34
Record Dates: First submitted 2022-11-30; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-06

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: virtual reality exposition — emotional response triggered by exposure to sensory stimuli presented in virtual reality.

SUMMARY:
Post-traumatic stress disorder (PTSD) develops after a threat for oneself and/or others. It is frequent, particularly in the military, due to repeated exposure to traumatic events. The prevalence is estimated between 35 and 75% in military.

It is essential to detect PTSD, whether it is present or sub-clinical, as early as possible, both from an individual point of view (maintaining the health of the soldier) and from a collective point of view (maintaining the operational status). Early detection is ²necessary for the implementation of early management strategies to reduce the significant risk of chronicization (around 80%), which can then be associated with severe complications such as addictions and suicide. The stakes of detecting PTSD are also at the collective level with the maintenance of operational capacity, under optimal performance and safety conditions (e.g.: risk of decompensation in the field with repercussions on the safety of the group and the progress of the mission).

However, the current methods of detecting PTSD (constituted or sub-clinical) is a clinical interview which can be associated with the use of the Clinical Administration PTSD for DSM -5 (CAPS) filled in by the clinician, or the self-reported questionnaires such as the Post-Traumatic CheckList Scale (PCL-5). It has many limitations, particularly due to the fear of stigmatization, which is greater in this professional context. Moreover, for sub-clinical PTSD, these tools are insufficient.

There is therefore a real need to develop screening tools for PTSD for soldiers that 1) are sensitive and specific (effectiveness), 2) are objective and do not depend on the answers given to a questionnaire (reliability), 3) can be implemented systematically on large samples (systematization), 4) do not depend on the soldier's spontaneous request for a health professional, and 5) are acceptable to the soldier (adherence). This need exists for constituted PTSD as well as for sub-clinical PTSD and constitutes a prerequisite for the implementation of early management (prevention of the risks of chronicization).

In view of the current data, PTSD can be considered as an emotional response (a conditioned fear response) because it is triggered in the absence of a real threat. To detect the presence or absence of PTSD, including sub-clinical PTSD, a proposition was made to characterize this emotional response triggered by exposure to sensory stimuli presented in virtual reality

DETAILED DESCRIPTION:
To develop and evaluate the robustness of a clinically constituted PTSD detection score (full PTSD) based on the emotional response, including conditioned fear, triggered by exposure to sensory stimuli presented in virtual reality and characterized by physiological and behavioral measures thus recorded

ELIGIBILITY:
Inclusion Criteria:

* military
* operational (fit to serve)
* men
* voluntary
* medical insurance

Exclusion Criteria:

* not military
* with medical or psychological suffering (other than PTSD or alcohol abuse)
* To develop and evaluate the robustness of a clinically constituted PTSD detection score
* not able to virtual reality

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The number of subjects needed per group is 20 or 80 subjects in total, to account for potential false negatives.
  This estimate is based on data from the few previous published studies using virtual reality to characterize the physiological responses of military personnel to various types of stimuli and thus to separate subjects (PTSD, sub-clinical PTSD and unaffected). The physiological measures used in our study are those from this literature (electrodermal conductance and heart rate) enriched with electroencephalographic recordings and behavioral biomarkers of interest because of their sensitivity described in the literature to emotional responses.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
physiological score for PTSD | one year
  To develop and evaluate the robustness of a clinically constituted PTSD detection score (full PTSD) based on the emotional response, including conditioned fear, triggered by exposure to sensory stimuli presented in virtual reality and characterized by physiological and behavioral measures thus recorded

SECONDARY OUTCOMES:
physiological score for partial PTSD | one year
  To evaluate and optimize the robustness of a clinically partial PTSD detection score

CONTACTS AND LOCATIONS:
Locations (1):
- DCSSA, Paris, Not in US/Canada, France

IPD SHARING:
Plan to Share IPD: Undecided
principal component analyses and algorithmy